CLINICAL TRIAL: NCT05746949
Title: Comparison of the Effects of High Flow Nasal Cannula Oxygen and Jet Ventilation Techniques on Oxygenation in Endolaryngeal Surgery: A Randomized Controlled Trial
Brief Title: Comparison of the Effects of High-flow Nasal Cannula Oxygen and Jet Ventilation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, attending anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/43
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Oxygen; pH; End-tidal Carbon Dioxide
Keywords: high-frequency jet ventilation; high flow nasal oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- jet ventilation group (No Intervention): Jet ventilation
- Optiflow group (Experimental): High flow nasal oxygen
  Interventions: Procedure: oxygenization techniques

INTERVENTIONS:
Procedure: oxygenization techniques — to compare the effects of high-flow nasal oxygen and jet ventilation on oxygenation in patients who will receive general anesthesia for endolaryngeal surgery.
  Arms: Optiflow group

SUMMARY:
Endoscopic microsurgical procedures of the larynx (direct examination-bx, microlaryngeal resection) require the anesthesiologist and surgeon to work in the same area throughout the procedure, and while ventilation is provided during the procedure, small diameter endotracheal tubes are preferred to see the surgical area as easily as possible.

However, it is sometimes observed that even conventional endotracheal tubes of this diameter make surgery difficult by obstructing the view. On the other hand, apneic laryngoscopy techniques used in upper airway surgeries, such as microlaryngoscopy and laryngotracheal surgery, where the airway is shared by the anesthesiologist and surgeon, have been replaced by safer and controlled high-frequency jet ventilation applications due to the risk of hypoxemia and hypercapnia.

In recent years, oxygenation has come to the fore with Transnasal High Flow Insufflation (OptiflowTM - Fischer & Paykel Healthcare, Auckland, New Zealand), an apneic oxygenation method.

This randomized study aimed to compare the effects of high-flow nasal oxygen and jet ventilation on oxygenation in patients receiving general anaesthesia for endolaryngeal surgery.

DETAILED DESCRIPTION:
Endoscopic microsurgical procedures of the larynx (direct examination- bx, microlaryngeal resection) require the anesthesiologist and surgeon to work in the same area throughout the procedure, and while ventilation is provided during the procedure, small diameter endotracheal tubes are preferred to see the surgical area as easily as possible.

However, it is sometimes observed that even conventional endotracheal tubes of this diameter make surgery difficult by obstructing the view.

On the other hand, apneic laryngoscopy techniques used in upper airway surgeries, such as microlaryngoscopy and laryngotracheal surgery, where the airway is shared by the anesthesiologist and surgeon, have been replaced by safer and controlled high-frequency jet ventilation applications due to the risk of hypoxemia and hypercapnia. In recent years, oxygenation has come to the fore with Transnasal High Flow Insufflation (OptiflowTM - Fischer & Paykel Healthcare, Auckland, New Zealand), an apneic oxygenation method. High-flow nasal cannula has been used, especially in critically ill patients. It is a system that delivers oxygen with high flow (up to 70 L/min) consisting of an air-oxygen mixer, an active heated humidifier, a single heated circuit and a nasal cannula.

Heated and humidified high-flow oxygen prolongs the time of preoxygenation and apneic oxygenation. In both jet ventilation and optiflow ventilation, gas exchange parameters of the patient can be measured by pulse oximetry, capnography, arterial blood gas or transcutaneous blood gas measurements. Determining the CO2 status (end-tidal CO2-ETCO2) in both techniques is quite difficult due to large leaks in the exhaled gas. Determining the patient's CO2 level is valuable as it shows the gas exchange. Ventilation settings are made according to this parameter. Arterial blood gas measurements can be performed for this purpose, but their invasiveness is limiting. An alternative method for assessing CO2 status is the nasal ETCO2 measurement. Evaluation of ventilation and oxygenation with nasally applied ETCO2 monitoring is a simple application that will bring patient safety to higher levels. In evaluating the adequacy of ventilation, basal ETCO2 values should be taken during the patients spontaneous breathing. This value should be compared with the values obtained during jet ventilation and transnasal high-flow oxygenation.

This randomized clinical study aims to compare the effects of high-flow nasal oxygen and jet ventilation on oxygenation in patients receiving general anaesthesia for endolaryngeal surgery.

After the approval of the Academic Ethics Committee, patients aged>18 years and ASA I-II,who are scheduled for endolaryngeal surgery under general anesthesia, will be included in the randomized study.

The patients will be randomized by the closed envelope method and divided into the jet ventilation group and the optiflow group. After premedication with midazolam 2mg IV, all patients will be taken to the operating room and monitored with standard monitoring methods (SPO2, KTA, SAB, DAB, OAB). In addition to standard monitoring, invasive arterial and nasal ETCO2 monitoring will be applied to all patients after general anesthesia induction. The patients in the first group will be ventilated with jet ventilation after induction, and the patients in the second group will be oxygenated with optiflow (OptiflowTM - Fischer & Paykel Healthcare, Auckland, New Zealand). Anesthesia will be maintained with remifentanil+propofol infusion in both groups. Anesthesia depth BIS (BIS PECTORAL INDEX) monitoring will be provided. At the end of the operation, all patients will be placed on conventional ventilation by placing a supraglottic airway, and decurarization will be provided with sugammadex. Arterial blood gas analysis will be recorded in all patients by measuring PaCO2, PaO2 and pH changes ( before induction, every 10 minutes after induction and at the end of the operation). During the operation, arterial blood gas was used as the primary output to record PaCO2 levels at five different times for all patients: before induction (T0) as baseline values, 10 minutes after induction (T1), 20 minutes after induction (T2), 30 minutes after induction (T3), and at the end of the operation (T4). As secondary outputs, arterial blood gas analysis recorded the patients' PaO2, pH, HCO3, BE, Hb, and lactate values, as well as vital parameters such as MAP, HR, and SpO2, at five separate times: before induction (T0) as baseline values, 10 minutes after induction (T1), 20 minutes after induction (T2), 30 minutes after induction (T3), and at the end of the operation (T4). Additionally, the highest PaO2 and PaCO2 values and the lowest SpO2 values during the perioperative period were recorded. Furthermore, the duration of the operation and changes in respiratory and hemodynamic parameters during the operation were evaluated.

This randomized study aimed to compare the effects of high-flow nasal oxygen and jet ventilation on oxygenation in patients who will receive general anesthesia for endolaryngeal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA I-II status
* Patients who will receive general anesthesia for endolaryngeal surgery
* >18 years old
* Volunteer to participate in the study

Exclusion Criteria:

* <18 years old
* MI (EF<%50)
* Arrhythmia
* Peripheral vascular disease
* Cerebrovascular disease
* Electrolyte disorder
* Severe COPD
* Chronic hypoxia
* BMI>35 kg/m2
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
PaCO2 change | Intraoperative
  PaCO2 change (before preoxygenation, before induction, every 5 minutes after induction) was recorded by arterial blood gas analysis.
Ph change | Intraoperative
  Ph changes (before preoxygenation, before induction, every 5 minutes after induction) were recorded by arterial blood gas analysis

SECONDARY OUTCOMES:
Arterial ETCO2 values | Intraoperative
  Arteryal ETCO2 values were evaluated with arterial blood gas and recorded.
Nasal ETCO2 values | Intraoperative
  Nasal ETCO2 values were evaluated with arterial blood gas and recorded.
Anesthesia duration | Intraoperative
  Anesthesia time was recorded
Surgery time | Intraoperative
  Surgery time was recorded
Surgical satisfaction questionnaire | Intraoperative
  Surgical satisfaction was evaluated and recorded
Respiratory complications | Intraoperative
  Possible respiratory complications were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Seda Özdağlı, Resident, Principal Investigator — Istanbul University; Demet Altun, Assoc. Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Lyons C, Callaghan M. Apnoeic oxygenation with high-flow nasal oxygen for laryngeal surgery: a case series. Anaesthesia. 2017 Nov;72(11):1379-1387. doi: 10.1111/anae.14036. PMID 29047136